CLINICAL TRIAL: NCT04381312
Title: COVID-19 Chez la Personne âgée de Plus de 70 Ans : Impact Direct et Indirect à 3 Mois.
Brief Title: Direct and Indirect Impact of COVID-19 In Older Populations
Acronym: COVID-OLD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC20.118; 2020-A00846-33 (Other: ID RCB)
Record Dates: First submitted 2020-04-10; First posted 2020-05-08 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2020-05

CONDITIONS: Risk Factors for COVID-19 Outcomes in Elderly Populations
Keywords: elderly; COVID 19; mortality; functional status
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study propose to describe risk factors for acute and long term mortality of COVID 19 in patients up to 70 years old.

DETAILED DESCRIPTION:
In December 2019, Wuhan city in China, became the center of an outbreak of pneumonia due to a novel coronavirus SARS-CoV-2, which disease was named coronavirus disease 2019 (COVID19) in February, 2020, by WHO. The COVID19 is much more dangerous for people over 60 with a death rate of 3.6% after 60, 8.0% after 70 and 14.8% after 80 -and according to our Italian colleagues over 20% after 90- against 2.3% in the general population. The elderly patients exhibits more complications (ARDS, delirium, cardiac and renal insufficiency) needing intensive care, and often had multiple comorbidities and in particular: cardiovascular disease (10.5% mortality), diabetes (7.3%), chronic respiratory disease (6.3%) and hypertension (6%).

Very few data are available the specific burden of Infectious diseases (ID) in older populations. The large majority of literature is often related to intrahospital or direct mortality and only recently arise the idea of indirect impact of ID particularly in that populations. In that meaning, ID may be considered as a trigger of other medical events such as myocardial infarction, stroke, or other specific outcomes such as functional decline; For the last 10 years, the Specific interest group " GInGer "( Groupe Infectio-Geriatrique ) a network of infectiologist and geriatrician SPILF/SFGG) carried out several studies on different aspects of ID in theses populations and recently demonstrated the indirect and long term impact of influenza and Clostridioides difficile infections. As an example, In influenza study, death-rate increases from 12,2 % in hospital related death to 25% at 3 months with high rate of complications (57%), high rates of rehospitalisation (25%) and functional decline (35%) leading to high increase in nursing home admission. The cost of these indirect impact is high and underestimated.

Because of incidence and comorbidities rates, severity of the actual French older COVID 19-infected older populations and because of the potential indirect and long term impact of COVID19 in these populations, it seems essential to know whether 3 month related death is largely higher as for influenza, to determine risk factors for intra hospital and long term death, measure acute and long term complications, and describe the impact of COVID 19 on specific ageing outcomes such as functional status at Month 3 (M3).

ELIGIBILITY:
Inclusion Criteria:

* + positive PCR confirmed COVID 19 (confirmed case) or positive Thoracic CT Scan - (probable case)

Exclusion Criteria:

* Direct admission in Intensive care.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Older populations admitted in acute care ward for COVID 19 eor in post acute care.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-04-09 (Actual); Primary Completion 2021-07-09 (Estimated); Study Completion 2021-10-09 (Estimated)

PRIMARY OUTCOMES:
mortality | 3 months
  3-month survival curve
Risk factors for death | 3 months
  Specific COVID 19 risk factors for death and geriatric risk factors for death
mortality | 12 months
  12 month survival curve
Risk factors for death | 12 months
  Specific COVID 19 risk factors for death and geriatric risk factors for death

SECONDARY OUTCOMES:
Describe clinical symptoms specific to old population | before and at admission
  clinical symptoms (respiratory , non respiratory symptoms and Geriatric syndromes)
describe specific and non-specific treatments used for COVID 19 | through study completion, an average of 1 year
  Prevalence and duration of specific treatments and non-specific treatments
describe all acute complications | through study completion, an average of 1 year
  prevalence of all medical usual complications and geriatric acquired complications, such as delirium, falls, complications, such as delirium, falls, malnutrition, pressure sore)
functional decline | 3 months post acute phase
  rates of Functional decline between basal status (before admission) and admission,and between basal and 3 months, and between Discharge and 3 month.
Rehospitalisation | 3 months post acute phase
  Prevalence of readmission to hospital
medical complications | 3 months post acute phase
  Prevalence of medical complication s ( new infectious disease, c cardiovascular, metabolic diseases and geriatric acquired complications, such as delirium, falls, complications, such as delirium, falls, malnutrition, pressure sore)
Admission in nursing home | 3 months post acute phase
  Prevalence of new nursing home admission
risk factors for 3-month functional decline, acute complication and admission to nursing home | 3 months post acute phase
  Determine risk factors for 3-month functional decline, acute complication and admission to nursing home

CONTACTS AND LOCATIONS:
Overall Officials: Gaetan GAVAZZI, Pr, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Chu Grenoble Alpes, Grenoble, Grenoble, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Background] Gavazzi G, Krause KH. Ageing and infection. Lancet Infect Dis. 2002 Nov;2(11):659-66. doi: 10.1016/s1473-3099(02)00437-1. PMID 12409046
- [Background] High KP, Bradley S, Loeb M, Palmer R, Quagliarello V, Yoshikawa T. A new paradigm for clinical investigation of infectious syndromes in older adults: assessment of functional status as a risk factor and outcome measure. Clin Infect Dis. 2005 Jan 1;40(1):114-22. doi: 10.1086/426082. Epub 2004 Dec 6. PMID 15614700
- [Background] Seynaeve D, Augusseau-Rivière B, Couturier P, Morel-Baccard C, Landelle C, Bosson JL, Gavazzi G, Mallaret MR. J Am Med Dir Assoc. 2019 May 14 Outbreak of human metapneumovirus in a French nursing home, a retrospective study? J Am Med Dir Assoc. 2019 May 14. pii: S1525-8610(19)30302-0. doi: 10.1016/j.jamda.2019.03.015
- [Background] Caupenne A, Ingrand P, Ingrand I, Forestier E, Roubaud-Baudron C, Gavazzi G, Paccalin M. Acute Clostridioides difficile Infection in Hospitalized Persons Aged 75 and Older: 30-Day Prognosis and Risk Factors for Mortality. J Am Med Dir Assoc. 2020 Jan;21(1):110-114. doi: 10.1016/j.jamda.2019.07.002. Epub 2019 Sep 17. PMID 31537480
- [Background] Gavazzi G, Paccalin M, de Wazieres B, Roubaud-Baudron C, Fraisse T, Bernard L, Legout L, Aquino JP, Guerin O, Forestier E, Burden of influenza in older patients over the 2016-2017 winter season in France. XXIXth ECCMID Amsterdam. (Nethderland) 2019